CLINICAL TRIAL: NCT00091182
Title: A Phase II Study of Oxaliplatin in Children With Recurrent Solid Tumors
Brief Title: Oxaliplatin in Treating Young Patients With Recurrent Solid Tumors That Have Not Responded to Previous Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01815; ADVL0421; COG-ADVL0421; CDR0000384560; U10CA098543 (NIH)
Record Dates: First submitted 2004-09-07; First posted 2004-09-09 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Childhood Central Nervous System Germ Cell Tumor; Childhood Extragonadal Germ Cell Tumor; Childhood Hepatoblastoma; Childhood Hepatocellular Carcinoma; Childhood High-grade Cerebral Astrocytoma; Childhood Low-grade Cerebral Astrocytoma; Childhood Malignant Ovarian Germ Cell Tumor; Childhood Malignant Testicular Germ Cell Tumor; Childhood Teratoma; Recurrent Adrenocortical Carcinoma; Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Ependymoma; Recurrent Childhood Liver Cancer; Recurrent Childhood Malignant Germ Cell Tumor; Recurrent Childhood Rhabdomyosarcoma; Recurrent Childhood Soft Tissue Sarcoma; Recurrent Childhood Visual Pathway and Hypothalamic Glioma; Recurrent Colon Cancer; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Nasopharyngeal Cancer; Recurrent Neuroblastoma; Recurrent Osteosarcoma; Recurrent Rectal Cancer; Recurrent Renal Cell Cancer
MeSH Terms: conditions — Hepatoblastoma; Astrocytoma; Ovarian Germ Cell Cancer; Testicular Neoplasms; Teratoma; Adrenocortical Carcinoma; Familial ependymoma; Optic Nerve Glioma; Colonic Neoplasms; Neuroectodermal Tumors, Primitive, Peripheral; Nasopharyngeal Neoplasms; Neuroblastoma; Osteosarcoma; Rectal Neoplasms; Carcinoma, Renal Cell | interventions — Oxaliplatin

ARMS (1):
- Arm I (Experimental): Patients receive oxaliplatin IV over 2 hours on day 1. Treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: oxaliplatin

INTERVENTIONS:
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP

SUMMARY:
This phase II trial is studying how well oxaliplatin works in treating young patients with recurrent solid tumors that have not responded to previous treatment. Drugs used in chemotherapy, such as oxaliplatin, work in different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the response rate in children with recurrent or refractory solid tumors treated with oxaliplatin.

II. Determine the cumulative toxicity of this drug in these patients. III. Determine the pharmacokinetic profile of this drug in these patients. IV. Determine time to progression and overall survival of patients treated with this drug.

V. Correlate the extent of oxaliplatin exposure with response in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to disease type.

Patients receive oxaliplatin IV over 2 hours on day 1. Treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed* solid tumor, including any of the following:

  * Ewing's sarcoma/peripheral primitive neuroectodermal tumor (PNET)
  * Osteosarcoma
  * Rhabdomyosarcoma
  * Neuroblastoma
  * High-grade astrocytoma
  * Low-grade astrocytoma
  * Glioblastoma multiforme
  * Ependymoma
  * Hepatoblastoma
  * Germ cell tumors of any site
  * Rare tumors of interest, including any of the following:

    * Soft tissue sarcoma
    * Hepatocellular carcinoma
    * Childhood/adolescent colorectal carcinoma
    * Childhood/adolescent renal cell carcinoma
    * Childhood/adolescent adrenocortical carcinoma
    * Childhood/adolescent nasopharyngeal carcinoma
* Recurrent disease OR refractory to conventional therapy
* Measurable disease by clinical exam, CT scan, MRI, or positron emission tomography
* Performance status - Karnofsky 50-100% (for patients over age 10)
* Performance status - Lansky 50-100% (for patients age 10 and under)
* At least 8 weeks
* Absolute neutrophil count ≥ 1,000/mm^3*
* Platelet count ≥ 75,000/mm^3* (transfusion independent)
* Hemoglobin ≥ 8.0 g/dL* (RBC transfusions allowed)
* Granulocytopenia, anemia, and/or thrombocytopenia due to bone marrow metastases or extensive prior radiotherapy allowed provided the above hematological criteria are met
* Bilirubin ≤ 3 mg/dL
* Creatinine based on age as follows:

  * ≤ .8 mg/dL (for patients age 5 and under)
  * ≤ 1.0 mg/dL (for patients age 6 to 10)
  * ≤ 1.2 mg/dL (for patients age 11 to 15)
  * ≤1.5 mg/dL (for patients age 16 to 21)
* Creatinine clearance or radioisotope glomerular filtration rate > 20 mL/min
* No uncontrolled seizure disorder
* No uncontrolled infection
* CNS toxicity ≤ grade 2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Recovered from prior immunotherapy
* At least 7 days since prior anticancer biologic therapy
* More than 1 week since prior growth factors
* At least 6 months since prior allogeneic stem cell transplantation

  * No evidence of active graft-vs-host disease
* No concurrent immunomodulating agents
* Recovered from prior chemotherapy
* No prior oxaliplatin
* Prior carboplatin or cisplatin allowed
* More than 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas)
* No other concurrent anticancer chemotherapy
* Concurrent dexamethasone for CNS tumors allowed provided patient has been on a stable or decreasing dose for ≥ 1 week before study entry
* Recovered from prior radiotherapy
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 6 months since prior craniospinal radiotherapy
* At least 6 months since prior radiotherapy to ≥ 50% of the pelvis
* At least 6 weeks since other prior substantial radiotherapy to the bone marrow
* Concurrent radiotherapy to localized painful lesions allowed provided ≥ 1 measurable lesion is not irradiated
* No other concurrent investigational agents
* No other concurrent anticancer agents

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Actual)
Dates: Start 2004-10; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 3 years
  Response rate and confidence intervals will be constructed according to the method of Chang and O'Brien.

CONTACTS AND LOCATIONS:
Overall Officials: Orren Beaty, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States